CLINICAL TRIAL: NCT04124497
Title: Daratumumab, Pomalidomide and Dexamethasone for Del(17p) Positive Relapsed and Relapsed/Refractory Multiple Myeloma Patients [DEDALO]
Brief Title: A Trial for Relapsed and Relapsed/Refractory Multiple Myeloma Patients
Acronym: DPd
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEDALO
Record Dates: First submitted 2019-07-02; First posted 2019-10-11 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma; Deletion 17P Syndrome
Keywords: Multiple Myeloma; Monoclonal antibody; Immunomodulating agents
MeSH Terms: conditions — Multiple Myeloma; Chromosome 17 deletion | interventions — daratumumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab Pomalidomide dexamethasone (Experimental): Therapy consists in cycles of the DPd combination as follows:
  * Pomalidomide 4 mg once daily on days 1-21;
  * Oral or intravenous dexamethasone 40 mg/day (≤ 75 years old) or 20 mg/ day (>75 years old) on days 1, 8, 15 and 22;
  * Daratumumab 16 mg/kg intravenously at following schedule:
  * cycle 1 and 2: days 1, 8, 15, and 22
  * cycle 3 through 6: days 1, and 15
  * from cycle 7 until disease progression: day 1.
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — * Daratumumab 16 mg/kg intravenously at following schedule:
  * cycle 1 and 2: days 1, 8, 15, and 22
  * cycle 3 through 6: days 1, and 15
  * from cycle 7 until disease progression: day 1.
  Other Names: Darzalex
Drug: Pomalidomide — 4 mg once daily on days 1-21
  Other Names: Imnovid
Drug: Dexamethasone — Oral or intravenous dexamethasone 40 mg/day (≤ 75 years old) or 20 mg/ day (>75 years old) on days 1, 8, 15 and 22

SUMMARY:
Multiple myeloma (MM) with chromosome 17 deletion (del(17p) represents one of the most dangerous genetic variant of this disease, since it is associated with a high level of genomic instability. Del(17p) is present in approximately 10% of patients at diagnosis, and its frequency increases with disease evolution. The adverse prognosis of del(17p) has been observed in patients treated with conventional chemotherapy and new drugs. Only very few studies have suggested an advantage in treating del(17p) MM patients with specific therapies. In particular, several recent trials combining lenalidomide plus dexamethasone with a new agent, suggested that high risk cytogenetics patients may benefit from newest generation drugs. Yet, in all studies, outcome of patients with high risk genetic features have been derived from subgroup analyses, with all the limitations of this approach. To date no trial has been designed with the specific aim to test genotype-adapted therapies.

The objective of the present study is to evaluate the combination of daratumumab-pomalidomide-dexamethasone (DPd) in relapsed or relapsed/refractory MM patients harboring del(17p).

Treatment of relapsed or relapsed/refractory MM patients harbouring del(17p) is a relevant unmet medical need. A clinical trial designed to test a tailored treatment for this patient population would be a major improvement. In this perspective the combination DPd seems attractive since:

* both daratumumab and pomalidomide are therapies not interfering with DNA replication, thus not increasing the intrinsic genomic instability of del(17p) plasma cells.
* the POLLUX study has shown that daratumumab in combination with lenalidomide is highly effective in relapsed and relapsed/refractory MM patients.10
* the IFM 2010-02 trial has suggested that pomalidomide may be effective in del(17p) patients.
* the DPd combination has been successfully tested in MM patients with advanced disease.

DETAILED DESCRIPTION:
Patients will undergo screening for protocol eligibility within 28 days (4 weeks) of enrolment.

After providing written informed consent to participate in the study, patients will be evaluated for study eligibility. It is to note that patients can be enrolled based on the presence of del(17p), as per center evaluation. However, the presence of del(17p) should be confirmed by the central laboratory (University of Torino laboratory), which will perform the test in 5 working days.

After registration, subjects who meet all the inclusion criteria will be treated according to the protocol, only after the presence of del(17p) has been confirmed by the central laboratory.

Treatment period includes administration of 28-day cycles of treatment with DPd until any sign of progression or intolerance.

The response will be assessed after each cycle. The LTFU period will start after development of confirmed progressive disease (PD) or treatment interruption due to toxicity. All patients are to be followed for survival during the LTFU period every 3 months via telephone or office visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given voluntary written informed consent
* Subject must be at least 18 years of age.
* Subject must have documented MM.
* Subject must have del(17p) observed by FISH in at least 10% of bone marrow plasma cells at any time of MM history.
* Subject must have serum monoclonal paraprotein (M-protein) level >=0.5 g/dL or urine M-protein, level >=200 mg/24 hours, or light chain MM, or serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* Subject must have received at least 1 and no more than 3 prior lines of therapy for MM.
* Subject must have received at least 2 consecutive cycles of lenalidomide in a previous line of therapy.
* Subject must have achieved a response (PR or better) to at least one prior regimen.
* Subjects must have either refractory or relapsed and refractory disease defined as documented disease progression during or within 60 days of completing their last myeloma therapy.
* Subject must have an ECOG Performance Status score of 0, 1, or 2.
* Subject must have the following laboratory values:

  * Platelet count >=50 x 109/L (≥30 x 109 /L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to drug administration).
  * Absolute neutrophil count (ANC) >= 1 x 109/L without the use of growth factors.
  * Corrected serum calcium <=14 mg/dL (3.5 mmol/L)
  * Alanine transaminase (ALT): <= 3 x the upper limit normal (ULN).
  * Total bilirubin: <= 2 x the ULN.
  * Calculated or measured creatinine clearance: >= 15 mL/minute
* Females of childbearing potential (FBCP) must follow the Pregnancy Prevention Plan and use a highly effective and an additional barrier contraception method simultaneously for 28 days before starting pomalidomide, during treatment and dose interruptions, for at least 28 days after the last dose of pomalidomide and 3 months after the last dose of daratumumab Males must use an effective barrier method of contraception if sexually active with FCBP for at least 28 days before starting pomalidomide, during the treatment and dose interruptions, for at least 28 days after the last dose of pomalidomide and 3 months after the last dose of daratumumab. Male subjects must agree to refrain from sperm donation for at least 3 months after the last dose of daratumumab.

Exclusion Criteria:

* Subject has received daratumumab or other anti-CD38 monoclonal antibody previously.
* Subject's disease shows evidence of refractoriness or intolerance to pomalidomide. If previously treated with a pomalidomide-containing regimen, the subject is excluded if he or she:

  * Discontinued due to any adverse event related to prior pomalidomide treatment, or
  * If, at any time point, the subject was refractory to any dose of pomalidomide.

Refractory to pomalidomide is defined either:

* Subjects whose disease progresses within 60 days of pomalidomide; or
* Subjects whose disease is nonresponsive while on lenalidomide. Nonresponsive disease is defined as either failure to achieve at least an MR or development of PD while on pomalidomide.

  * Subject has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the date of randomization.
  * Subjects who received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant less than 12 months prior to initiation of study treatment and who have not discontinued immunosuppressive treatment for at least 16 weeks prior to initiation of study treatment and are currently dependent on such treatment.
  * Subjects unable or unwilling to undergo antithrombotic prophylactic treatment.
  * Subject has a history of malignancy (other than multiple myeloma) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, in agreement with the medical monitor, is considered cured with minimal risk of recurrence within 3 years).
  * Subject has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume in 1 second (FEV1) <60% of predicted normal), asthma, or a history of asthma within the last 2 years. Subjects with known or suspected COPD must have a forced expiratory volume (FEV) test during Screening.
  * Subject is known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg] or antibodies to hepatitis B surface and core antigens [anti-HBs and anti-HBc, respectively]) or hepatitis C (anti-HCV antibody positive or HCV-RNA quantitation positive).
  * Subject has any concurrent medical condition or disease (eg, active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
  * Subject has clinically significant cardiac disease, including:
* Myocardial infarction within 6 months before Cycle 1, Day 1, or unstable or
* uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV)
* Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] Version 4 Grade 2 or higher) or clinically significant ECG abnormalities.
* Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >500 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) | 5 years
  Molecular minimal residual disease (MRD) 10-5 negativity rate assessed by means of next-generation sequencing (ClonoSEQ assay) in patients attaining a complete remission in the first year of treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 years
  Number of months from the date of randomization to the date of first observation of PD, or death from any cause as an event.
Overall response rate (ORR) | 5 years
  Overall response rate will include complete response (CR), very good partial response (VGPR) and partial response (PR) using the International Response Criteria. Responders are defined as subjects with at least a PR.
Progression-free survival 2 (PFS2) | 5 years
  Time from randomization to objective tumor progression on next-line treatment or death from any cause.
Duration of response (DOR) | 5 years
  Time between first documentation of response and PD. Responders without disease progression will be censored either at the time of lost to FU, at the time of death due to other cause than PD, or at the end of the study.
Overall survival (OS) | 5 years
  Time between randomization and death. Subjects who die will be censored at time of death as an event, regardless cause of death.
Safety as incidence of toxicities | 5 years
  Severity of the toxicities will be graded according to the NCI CTC v.5 whenever possible. Laboratory data will be graded according to NCI CTC v.5 severity grade.
Time to next therapy (TNT) | 5 years
  Time to next therapy will be measured from the date of randomization to the date of next anti-myeloma therapy. Death due to any cause before starting therapy will be considered an event.
Percentage of patients with negative MRD and survival indices | 5 years
  MRD negativity rate and survival might significantly change in particular subgroups of patients, that are defined on prognostic factors [ISS stage, additional cytogenetic abnormalities, previous treatment, presence of del(17p)]. Hence, subgroup analyses will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Montefusco, Principal Investigator — Ospedale San Carlo Borromeo - Italy
Locations (15):
- Italy (15):
  - AOU Ospedali Riuniti Umberto I, Ancona
  - Policlinico-Università degli Studi, Bari
  - Ospedali Riuniti, Bergamo
  - Policlinico S. Orsola, Bologna
  - A.O. Spedali Civili di Brescia, Brescia
  - AOU Policlinico Vittorio Emanuele, Catania
  - Ospedale Niguarda Cà Grande, Milan
  - Ospedale Maggiore, Novara
  - Dipart. Di Medicina Interna e Scienze Biomediche, Parma
  - Ospedale Oncologico Regionale, Rionero in Vulture
  - Policlinico Umberto I - Università La Sapienza, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.O. Santa Maria, Terni
  - AOU Città della Salute e della Scienza di Torino - Presidio Molinette, Torino
  - Policlinico Universitario di Udine, Udine

IPD SHARING:
Plan to Share IPD: No